CLINICAL TRIAL: NCT06065241
Title: Randomized Double Blind Placebo-controlled Trial to Investigate the Effect of a Botanical Formulation, LLP-01, on Proteomic Inflammatory and Cardiovascular Biomarkers.
Brief Title: Quantifiably Determine if the Botanical Formulation, LLP-01, Has a Significant Clinical Effect on Proteomic Inflammatory and Cardiovascular Biomarkers in Healthy, Older Individuals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LL Prosper Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SDLLP-01
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Aging; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: 2 month, double blind placebo controlled study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in this arm will receive a herbal capsule formulation, called LLP-01, consisting of 2 capsules taken once daily without food for 60 days. The capsules contain extracts from naturally occurring plant species, including Withania somnifera, Rosmarinus officinalis, Curcuma longa, Cotinus coggygria, Panax ginseng, Cordyceps militaris, Camellia sinensis, Cotinus coggygria, and Piper nigrum.
  Interventions: Dietary Supplement: LLP-01
- Placebo Group (Placebo Comparator): Participants in this arm will receive Placebo capsules, which are visually identical to the capsules in the Experimental Group. These placebo capsules are filled with rice flour and a minor amount of Curcuma longa powder and should be taken in the same manner as the Experimental Group, with 2 capsules taken once daily without food for 60 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: LLP-01 — Participants in the experimental group will take 2 capsules daily containing 1,000mg of the formulation, LLP-01, for 60 days.
  Arms: Experimental Group
Other: Placebo — Participants in the placebo group will take 2 capsules daily containing rice flower and small amount of Curcuma Longa for 60 days.
  Arms: Placebo Group

SUMMARY:
This is a prospective, interventional, double-blinded placebo-controlled study of up to 40 participants to evaluate the effect of a botanical formulation on inflammatory and cardiovascular biomarkers .

DETAILED DESCRIPTION:
The objective of this study is to understand the impact of a multi-botanical formulation on measurements of protein markers, with a focus on inflammation over a 60-day period. The primary objective of this study is to assess the effect of the formulation, LLP-01, on inflammatory and cardiovascular proteomic biomarkers. Adverse events will be self-monitored by participants and will be reported. Changes in weight/calculated BMI and grip strength, as well as changes in well-being through a self-reported questionnaire will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-75 years of age
* Any sex / gender
* All ethnicities
* Able to participate in a 2 month trial
* Able to provide informed consent
* Participant must be able to comply with treatment plan and laboratory tests
* Can swallow 00 size capsules

Exclusion Criteria:

* Any clinically diagnosed medical disease or disorder that requires prescribed medication(s)
* Currently on any anticoagulant medicines, such as warfarin
* Planned surgical procedure during study period
* Consumption of any supplements within the last 30 days that include the following botanicals/ingredients: green tea extract, Ashwagandha, Fisetin, Curcumin/Turmeric extract, Rosemary extract, Cordyceps, Ginseng
* Allergy or other sensitivity to any of the botanicals in the investigated product
* Currently or have been sick (bacterial or viral infection) in the last 14 days
* Alcoholism or drug addiction
* Participation in a clinical research trial within 30 days prior to enrollment in this trial
* Cognitive impairment, illiteracy, inability or unwillingness to give voluntary informed consent
* Unable or unwilling to provide required blood sample for testing and for use in a scientific publication (personal information undisclosed)
* Participants with any condition that may preclude venipuncture/ venous blood draw

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Plasma Proteomic Changes | Change from baseline to 60 days and compared to placebo
  Serum proteomic test to measure significant effects on any of the plasma proteins that will be analyzed. These proteins represent inflammatory, and cardiovascular responses, as well as metabolic functions.

SECONDARY OUTCOMES:
Grip Strength | Change from baseline to 60 days and compared to placebo
  Digital grip strength device to measure absolute grip strength
Weight/BMI | Change from baseline to 60 days and compared to placebo
  Height and weight to measuring absolute weight and to calculate BMI
Well-being | Change from baseline to 60 days and compared to placebo
  Questionnaire covering different aspects of well-being

CONTACTS AND LOCATIONS:
Overall Officials: Adi Ramon, M.Sc, Principal Investigator — Chief Compliance Officer
Locations (1):
- LL Prosper Inc., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided